CLINICAL TRIAL: NCT00676650
Title: A Multicenter, Randomized, Double-Blind, Phase 3 Study Of Sunitinib Plus Prednisone Versus Prednisone In Patients With Progressive Metastatic Castration-Resistant Prostate Cancer After Failure Of A Docetaxel-Based Chemotherapy Regimen
Brief Title: Sunitinib Plus Prednisone In Patients With Metastatic Castration-Resistant Prostate Cancer After Failure Of Docetaxel Chemotherapy
Acronym: SUN 1120
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study A6181120 was prematurely discontinued due to futility on 27 September 2010. No new or unexpected safety issues were identified.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A6181120
Record Dates: First submitted 2008-05-08; First posted 2008-05-13 (Estimated); Results first posted 2013-03-08 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2013-02

CONDITIONS: Prostatic Neoplasms
Keywords: Docetaxel-refractory mCRPC; Second-line treatment with sunitinib and prednisone
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Prednisone; Sunitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Treatment Arm A - sunitinib + prednisone
  Interventions: Drug: Prednisone; Drug: sunitinib
- B (Placebo Comparator): Treatment Arm B - placebo + prednisone
  Interventions: Drug: Placebo; Drug: Prednisone

INTERVENTIONS:
Drug: Prednisone — 5 mg BID, oral
  Other Names: Deltasone
  Arms: A
Drug: sunitinib — 37.5 mg/day, oral, administered on a continuous daily dosing regimen
  Other Names: Sutent, SU011248
  Arms: A
Drug: Placebo — 37.5 mg/day, oral, administered on a continuous daily dosing regimen
  Arms: B
Drug: Prednisone — 5 mg BID, oral
  Other Names: Deltasone
  Arms: B

SUMMARY:
This study will compare the safety and efficacy of sunitinib in combination with prednisone versus placebo and prednisone in patients that have metastatic castration-resistant prostate cancer that has progressed after treatment with a docetaxel-containing chemotherapy regimen. This is a second-line study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate.
* Progressive, metastatic castration-resistant prostate cancer after failure of docetaxel chemotherapy (resistant or intolerant).
* Progressive disease based on PSA progression, RECIST, or positive bone scan.
* ECOG 0 or 1.

Exclusion Criteria:

* Prior treatment with sunitinib and/or more than 1 prior chemotherapy regimen in the metastatic disease setting.
* Chemotherapy within 3 weeks.
* Impending complications from bone metastases.
* Ongoing urinary obstruction.
* Cardiac dysfunction, QTc >470 msec.
* CNS involvement.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 873 (Actual)
Dates: Start 2008-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (182):
- United States (76):
  - Pfizer Investigational Site, Decatur, Alabama
  - Pfizer Investigational Site, Huntsville, Alabama
  - Pfizer Investigational Site, Anaheim, California
  - Pfizer Investigational Site, Encinitas, California
  - Pfizer Investigational Site, Glendale, California
  - Pfizer Investigational Site, La Jolla, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Modesto, California
  - Pfizer Investigational Site, Thousand Oaks, California
  - Pfizer Investigational Site, Thousands Oaks, California
  - Pfizer Investigational Site, Vista, California
  - Pfizer Investigational Site, Westlake Village, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Lafayette, Colorado
  - Pfizer Investigational Site, Gainesville, Florida
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Winter Park, Florida
  - Pfizer Investigational Site, Arlington Heights, Illinois
  - Pfizer Investigational Site, Niles, Illinois
  - Pfizer Investigational Site, Winfield, Illinois
  - Pfizer Investigational Site, Zion, Illinois
  - Pfizer Investigational Site, Carmel, Indiana
  - Pfizer Investigational Site, Fishers, Indiana
  - Pfizer Investigational Site, Greenfield, Indiana
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Lafayette, Indiana
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Danvers, Massachusetts
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, Saint Cloud, Minnesota
  - Pfizer Investigational Site, Corinth, Mississippi
  - Pfizer Investigational Site, Southaven, Mississippi
  - Pfizer Investigational Site, Lincoln, Nebraska
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Henderson, Nevada
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Sewell, New Jersey
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, The Bronx, New York
  - Pfizer Investigational Site, Cary, North Carolina
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Kernersville, North Carolina
  - Pfizer Investigational Site, Lexington, North Carolina
  - Pfizer Investigational Site, Mount Airy, North Carolina
  - Pfizer Investigational Site, North Wilkesboro, North Carolina
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Bismarck, North Dakota
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Mayfield Heights, Ohio
  - Pfizer Investigational Site, Mentor, Ohio
  - Pfizer Investigational Site, Orange, Ohio
  - Pfizer Investigational Site, Westlake, Ohio
  - Pfizer Investigational Site, Eugene, Oregon
  - Pfizer Investigational Site, Springfield, Oregon
  - Pfizer Investigational Site, Clairton, Pennsylvania
  - Pfizer Investigational Site, Greensburg, Pennsylvania
  - Pfizer Investigational Site, Johnstown, Pennsylvania
  - Pfizer Investigational Site, Kingston, Pennsylvania
  - Pfizer Investigational Site, Lancaster, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Uniontown, Pennsylvania
  - Pfizer Investigational Site, Wexford, Pennsylvania
  - Pfizer Investigational Site, Brighton, Tennessee
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Arlington, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Fort Worth, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Webster, Texas
  - Pfizer Investigational Site, Everett, Washington
  - Pfizer Investigational Site, Monroe, Washington
  - Pfizer Investigational Site, Seattle, Washington
  - Pfizer Investigational Site, Milwaukee, Wisconsin
- Australia (4):
  - Pfizer Investigational Site, Port Macquarie, New South Wales
  - Pfizer Investigational Site, Wahroong, New South Wales
  - Pfizer Investigational Site, Westmead, New South Wales
  - Pfizer Investigational Site, Wodonga, Victoria
- Belgium (5):
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Liège
  - Pfizer Investigational Site, Mons
  - Pfizer Investigational Site, Namur
  - Pfizer Investigational Site, Wilrijk
- Brazil (6):
  - Pfizer Investigational Site, Salvador, Estado de Bahia
  - Pfizer Investigational Site, Belo Horizonte, Minas Gerais
  - Pfizer Investigational Site, Rio de Janeiro, Rio de Janeiro
  - Pfizer Investigational Site, Caxias do Sul, Rio Grande do Sul
  - Pfizer Investigational Site, Porto Alegre, Rio Grande do Sul
  - Pfizer Investigational Site, Santo André, São Paulo
- Canada (5):
  - Pfizer Investigational Site, Kelowna, British Columbia
  - Pfizer Investigational Site, Barrie, Ontario
  - Pfizer Investigational Site, Oshawa, Ontario
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Sherbrooke, Quebec
- China (4):
  - Pfizer Investigational Site, Wuhan, Hubei
  - Pfizer Investigational Site, Beijing
  - Pfizer Investigational Site, Chongqing
  - Pfizer Investigational Site, Shanghai
- Czechia (3):
  - Pfizer Investigational Site, Brno
  - Pfizer Investigational Site, Olomouc
  - Pfizer Investigational Site, Ústí nad Labem
- Denmark (4):
  - Pfizer Investigational Site, Herlev
  - Pfizer Investigational Site, Koebenhavn Oe
  - Pfizer Investigational Site, Odense C
  - Pfizer Investigational Site, Vejle
- Finland (2):
  - Pfizer Investigational Site, Helsinki
  - Pfizer Investigational Site, Tampere
- France (11):
  - Pfizer Investigational Site, Besançon
  - Pfizer Investigational Site, Bordeaux
  - Pfizer Investigational Site, Clermont-Ferrand
  - Pfizer Investigational Site, Lille
  - Pfizer Investigational Site, Lyon
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Poitiers
  - Pfizer Investigational Site, Rennes
  - Pfizer Investigational Site, Rouen
  - Pfizer Investigational Site, Saint-Grégoire
  - Pfizer Investigational Site, Tours
- Germany (8):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Homburg/Saar
  - Pfizer Investigational Site, Kempen
  - Pfizer Investigational Site, Leipzig
  - Pfizer Investigational Site, München
  - Pfizer Investigational Site, Münster
  - Pfizer Investigational Site, Tübingen
  - Pfizer Investigational Site, Ulm
- Israel (4):
  - Pfizer Investigational Site, Kfar Saba
  - Pfizer Investigational Site, Petah Tikva
  - Pfizer Investigational Site, Tel Litwinsky
  - Pfizer Investigational Site, Ẕerifin
- Italy (8):
  - Pfizer Investigational Site, Meldola, FC
  - Pfizer Investigational Site, Lido Di Camaiore (LU)
  - Pfizer Investigational Site, Napoli
  - Pfizer Investigational Site, Padua
  - Pfizer Investigational Site, Pavia
  - Pfizer Investigational Site, Pisa
  - Pfizer Investigational Site, Potenza
  - Pfizer Investigational Site, Roma
- Peru (3):
  - Pfizer Investigational Site, Arequipa, Arequipa
  - Pfizer Investigational Site, Lima, Lima Province
  - Pfizer Investigational Site, Bellavista, Provincia Constitucional del Callao
- Poland (3):
  - Pfizer Investigational Site, Gdansk
  - Pfizer Investigational Site, Kielce
  - Pfizer Investigational Site, Warsaw
- Portugal (2):
  - Pfizer Investigational Site, Porto
  - Pfizer Investigational Site, Setúbal
- Slovakia (4):
  - Pfizer Investigational Site, Bratislava
  - Pfizer Investigational Site, Martin
  - Pfizer Investigational Site, Prešov
  - Pfizer Investigational Site, Žilina
- South Korea (3):
  - Pfizer Investigational Site, Goyang-si, Gyeonggi-do
  - Pfizer Investigational Site, Seongnam, Gyunggido
  - Pfizer Investigational Site, Seoul
- Spain (10):
  - Pfizer Investigational Site, A Coruña, A Coruña
  - Pfizer Investigational Site, Elche, Alicante
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, L'Hospitalet de Llobregat, Barcelona
  - Pfizer Investigational Site, Girona, Gerona
  - Pfizer Investigational Site, Guadalajara, Guadalajara
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Pamplona, Navarre
  - Pfizer Investigational Site, Seville, Sevilla
  - Pfizer Investigational Site, Valencia, Valencia
- Sweden (4):
  - Pfizer Investigational Site, Lund
  - Pfizer Investigational Site, Malmo
  - Pfizer Investigational Site, Stockholm
  - Pfizer Investigational Site, Vaxjo
- Taiwan (3):
  - Pfizer Investigational Site, Taichung
  - Pfizer Investigational Site, Taipei
  - Pfizer Investigational Site, Taoyuan District
- United Kingdom (10):
  - Pfizer Investigational Site, Bournemouth, Dorset
  - Pfizer Investigational Site, Preston, Lancashire
  - Pfizer Investigational Site, Northwood, Middlesex
  - Pfizer Investigational Site, Bristol
  - Pfizer Investigational Site, Cardiff
  - Pfizer Investigational Site, Glasgow
  - Pfizer Investigational Site, Guildford
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Sheffield
  - Pfizer Investigational Site, Swansea

REFERENCES:
- [Derived] Michaelson MD, Oudard S, Ou YC, Sengelov L, Saad F, Houede N, Ostler P, Stenzl A, Daugaard G, Jones R, Laestadius F, Ullen A, Bahl A, Castellano D, Gschwend J, Maurina T, Chow Maneval E, Wang SL, Lechuga MJ, Paolini J, Chen I. Randomized, placebo-controlled, phase III trial of sunitinib plus prednisone versus prednisone alone in progressive, metastatic, castration-resistant prostate cancer. J Clin Oncol. 2014 Jan 10;32(2):76-82. doi: 10.1200/JCO.2012.48.5268. Epub 2013 Dec 9. PMID 24323035
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181120&StudyName=Sunitinib%20Plus%20Prednisone%20In%20Patients%20With%20Metastatic%20Castration-Resistant%20Prostate%20Cancer%20After%20Failure%20Of%20Docetaxel%20Chemotherapy

RESULTS

PARTICIPANT FLOW:
Groups:
- Sunitinib and Prednisone: Sunitinib capsules administered orally as a continuous daily dose in a continuous regimen, expressed as 4-week cycles; starting dose of 37.5 milligrams (mg) with option to increase dose to 50 mg at Cycle 3. Prednisone administered continuously at 5 mg orally twice a day (BID) as either a tablet, solution or concentrated solution.
- Placebo and Prednisone: Matched placebo administered orally as a continuous daily dose expressed as 4-week cycles; with a starting dose of 37.5 milligrams (mg) with option to increase dose to 50 mg at Cycle 3 plus prednisone administered continuously at 5 mg orally BID as either a tablet, solution or concentrated solution.
Period: Overall Study
Arm/Group | Sunitinib and Prednisone | Placebo and Prednisone
Started | 584 | 289
Treated | 581 | 285
Completed | 0 | 0
Not Completed | 584 | 289
Not completed — Death | 45 | 14
Not completed — Adverse Event | 159 | 21
Not completed — Global deterioration of health status | 66 | 31
Not completed — Lost to Follow-up | 0 | 1
Not completed — Objective progression or relapse | 189 | 140
Not completed — Other | 14 | 10
Not completed — Protocol Violation | 3 | 1
Not completed — Study terminated by sponsor | 57 | 43
Not completed — Withdrawal by Subject | 48 | 24
Not completed — Randomized but not treated | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sunitinib and Prednisone | Placebo and Prednisone | Total
Number analyzed (Participants) | 584 | 289 | 873
Age, Customized [Number; unit: participants]
  18 - 44 years | 3 | 0 | 3
  45 - 64 years | 177 | 97 | 274
  greater than or equal to (>=) 65 years | 404 | 192 | 596
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 584 | 289 | 873

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS is the duration from randomization to death. For participants who were alive, overall survival was censored at the last contact. OS (in months) calculated as (date of death minus [-] date of randomization plus [+] 1) divided (/) 30.4.
Time Frame: Baseline up to 32 months
Population: Full analysis (FA) population: all participants who were randomized, with study drug assignment designated according to initial randomization, regaradless of whether participant received study drug according to the randomization schedule.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sunitinib and Prednisone | Placebo and Prednisone
Number analyzed (Participants) | 584 | 289
months | 13.1 [12.0 to 14.1] | 11.8 [10.8 to 14.2]
Statistical Analysis 1: Comparison: Sunitinib and Prednisone vs Placebo and Prednisone; Test type: Superiority or Other; p = 0.1678, Log Rank — 1-sided p-value from the stratified log-rank test; Hazard Ratio (HR) = 0.914, 95% CI 2-sided [0.762 to 1.097] — Based on the Cox Proportional hazards model stratified by Eastern Cooperative Oncology Group (ECOG) and Disease Progression Base

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS is the period from randomization until disease progression or death on study. PFS is censored on the date of last tumor assessment documenting absence of progressive disease. PFS (weeks) calculated as (first event date - randomization date + 1)/7.02
Time Frame: Baseline, every 8 weeks up to 123 weeks
Population: FA Population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Sunitinib and Prednisone | Placebo and Prednisone
Number analyzed (Participants) | 584 | 289
weeks | 24.1 [23.4 to 28.1] | 17.9 [15.8 to 24.1]
Statistical Analysis 1: Comparison: Sunitinib and Prednisone vs Placebo and Prednisone; Test type: Superiority or Other; p < 0.001, Log Rank — 1-sided p-value from the stratified log-rank test; Hazard Ratio (HR) = 0.725, 95% CI 2-sided [0.591 to 0.890] — Based on Cox Proportional Hazards Model stratified by ECOG and Disease Progression Base

3. Secondary Outcome: Percent of Participants With Objective Response (OR)
Description: OR defined as the percent (%) of participants with confirmed Complete Response (CR) (disappearance of all target lesions) or Partial Response (PR) (>=30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions) according to Response Evaluation Criteria in Solid Tumors (RECIST), relative to the full analysis population. Confirmed responses were those that persist on repeat imagining study >= 4 weeks after initial documentation of response.
Time Frame: Baseline, every 8 weeks up to 123 weeks
Population: FA Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sunitinib and Prednisone | Placebo and Prednisone
Number analyzed (Participants) | 584 | 289
percentage of participants | 6.1 [3.8 to 9.3] | 1.8 [0.4 to 5.2]
Statistical Analysis 1: Comparison: Sunitinib and Prednisone vs Placebo and Prednisone; Test type: Superiority or Other; p = 0.040, Fisher Exact — p-value from 2-sided Fisher's Exact test; Odds Ratio (OR) = 3.561, 95% CI 2-sided [1.0 to 19.0]

4. Secondary Outcome: Duration of Response (DR)
Description: Time in weeks from the first documentation of objective tumor response to objective tumor progression or death due to any cause. Duration of tumor response was calculated as (the date of the first documentation of objective tumor progression or death due to cause - the date of the first CR or PR that was subsequently confirmed plus 1 divided by 7.02. DR calculated for the subgroup of participants with a confirmed objective tumor response
Time Frame: Baseline, every 8 weeks up to 123 weeks
Population: Data not summarized, study terminated early
Arm/Group | Sunitinib and Prednisone | Placebo and Prednisone
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change From Baseline in Pain Severity
Description: Pain severity recorded on a numerical scale ranging from 0 (no pain) to 10 (pain as bad as you can imagine). Higher scores indicated greater level of pain. The pain score for each cycle averaged for the 7 days.
Time Frame: Day 1 through Day 7 every 28 days (every cycle) up to 29 months
Population: Data not summarized, study terminated early
Arm/Group | Sunitinib and Prednisone | Placebo and Prednisone
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy-Prostate (FACT-P)
Description: FACT-P is a validated, self-administered instrument used to assess health-related quality of life and prostate cancer-specific symptoms. Scores ranged from 0 (not at all) to 4 (very much). It is 27-item FACT-General and 12 items for the prostate cancer specific concerns. The 27 items in FACT-G are grouped into 4 domains: physical well-being, social/family well-being, emotional well-being and functional well-being. The 12 prostate cancer symptoms items focus on pain (3 items), urination problems (3 items), sexual functions (2 items), weight loss, appetite, overall comfort, and bowel movement.
Time Frame: Baseline, every 4 weeks up to 123 weeks
Population: Data not summarized, study terminated early
Arm/Group | Sunitinib and Prednisone | Placebo and Prednisone
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change From Baseline in Euro Quality of Life (EQ-5D)- Health State Profile Utility Score
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state ("confined to bed"). Overall scores range from 0 to 1, with lower scores representing a higher level of dysfunction.
Time Frame: Baseline, every 4 weeks up to 123 weeks
Population: Data not summarized, study terminated early
Arm/Group | Sunitinib and Prednisone | Placebo and Prednisone
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Sunitinib and Prednisone | Placebo and Prednisone
Serious Adverse Events (participants affected / at risk) | 275/581 | 86/285
Other Adverse Events (participants affected / at risk) | 573/581 | 256/285
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib and Prednisone (N=581) | Placebo and Prednisone (N=285)
Anaemia (Blood and lymphatic system disorders) | 21 | 3
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 1
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0
Leukopenia (Blood and lymphatic system disorders) | 3 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 3 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 1
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 3 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 2 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 2 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Cerebral arteriovenous malformation haemorrhagic (Congenital, familial and genetic disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Vestibular disorder (Ear and labyrinth disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 1
Conjunctival oedema (Eye disorders) | 1 | 0
Diplopia (Eye disorders) | 1 | 0
Optic ischaemic neuropathy (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Anal fistula (Gastrointestinal disorders) | 2 | 0
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0
Anal ulcer (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 3
Diarrhoea (Gastrointestinal disorders) | 7 | 1
Diverticular perforation (Gastrointestinal disorders) | 1 | 0
Duodenitis (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 4 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 7 | 1
Gingival bleeding (Gastrointestinal disorders) | 2 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Large intestine perforation (Gastrointestinal disorders) | 2 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 3 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 13 | 4
Oesophagitis (Gastrointestinal disorders) | 3 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Peptic ulcer (Gastrointestinal disorders) | 1 | 0
Proctitis (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 1
Rectal ulcer (Gastrointestinal disorders) | 2 | 0
Rectal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Rectourethral fistula (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 16 | 5
Asthenia (General disorders) | 14 | 1
Chest pain (General disorders) | 3 | 2
Death (General disorders) | 5 | 1
Device occlusion (General disorders) | 2 | 1
Disease progression (General disorders) | 32 | 19
Fatigue (General disorders) | 2 | 1
General physical health deterioration (General disorders) | 10 | 2
Ill-defined disorder (General disorders) | 2 | 0
Impaired healing (General disorders) | 1 | 0
Influenza like illness (General disorders) | 1 | 0
Malaise (General disorders) | 2 | 0
Medical device complication (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 2 | 0
Pain (General disorders) | 2 | 4
Performance status decreased (General disorders) | 2 | 0
Pyrexia (General disorders) | 11 | 3
Sudden cardiac death (General disorders) | 1 | 0
Sudden death (General disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 4 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Gallbladder disorder (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 1
Hepatitis cholestatic (Hepatobiliary disorders) | 1 | 0
Hepatorenal failure (Hepatobiliary disorders) | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Anal abscess (Infections and infestations) | 6 | 0
Appendicitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Cholecystitis infective (Infections and infestations) | 1 | 0
Clostridial infection (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 4 | 0
Febrile infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 0
Herpes zoster (Infections and infestations) | 1 | 1
Infection (Infections and infestations) | 4 | 0
Infectious peritonitis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Meningitis bacterial (Infections and infestations) | 0 | 1
Oral fungal infection (Infections and infestations) | 1 | 0
Otitis media chronic (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 0 | 1
Perirectal abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 4 | 4
Pseudomonas infection (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Rectal abscess (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 3 | 0
Septic shock (Infections and infestations) | 2 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 10 | 7
Urinary tract infection bacterial (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 1 | 1
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Cystitis radiation (Injury, poisoning and procedural complications) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 5 | 1
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 2 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 2 | 0
Blood urea increased (Investigations) | 2 | 0
C-reactive protein increased (Investigations) | 0 | 1
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 2 | 0
Prothrombin time prolonged (Investigations) | 1 | 0
Urine output decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 6 | 2
Dehydration (Metabolism and nutrition disorders) | 17 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 10 | 5
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Aphasia (Nervous system disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 3 | 0
Convulsion (Nervous system disorders) | 2 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 3 | 0
Facial paresis (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 1 | 0
Hydrocephalus (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 2 | 0
Nervous system disorder (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 2 | 0
Partial seizures (Nervous system disorders) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Polyneuropathy in malignant disease (Nervous system disorders) | 0 | 1
Post herpetic neuralgia (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 3 | 3
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 3 | 0
Transient ischaemic attack (Nervous system disorders) | 2 | 0
VIIth nerve paralysis (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 3 | 3
Hallucination (Psychiatric disorders) | 1 | 0
Mental disorder due to a general medical condition (Psychiatric disorders) | 2 | 0
Azotaemia (Renal and urinary disorders) | 1 | 0
Bladder obstruction (Renal and urinary disorders) | 1 | 0
Bladder tamponade (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 1
Haematuria (Renal and urinary disorders) | 13 | 3
Hydronephrosis (Renal and urinary disorders) | 1 | 2
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0
Obstructive uropathy (Renal and urinary disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 1 | 1
Renal failure acute (Renal and urinary disorders) | 8 | 2
Renal impairment (Renal and urinary disorders) | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 2 | 0
Urethral haemorrhage (Renal and urinary disorders) | 1 | 0
Urinary bladder haemorrhage (Renal and urinary disorders) | 3 | 0
Urinary retention (Renal and urinary disorders) | 3 | 3
Urinary tract obstruction (Renal and urinary disorders) | 1 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 19 | 3
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Pain management (Surgical and medical procedures) | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 4 | 1
Haematoma (Vascular disorders) | 1 | 0
Haemorrhage (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 4 | 0
Hypotension (Vascular disorders) | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib and Prednisone (N=581) | Placebo and Prednisone (N=285)
Anaemia (Blood and lymphatic system disorders) | 140 | 53
Leukopenia (Blood and lymphatic system disorders) | 60 | 2
Neutropenia (Blood and lymphatic system disorders) | 84 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 72 | 8
Abdominal pain (Gastrointestinal disorders) | 41 | 13
Abdominal pain upper (Gastrointestinal disorders) | 39 | 10
Constipation (Gastrointestinal disorders) | 112 | 56
Diarrhoea (Gastrointestinal disorders) | 267 | 43
Dry mouth (Gastrointestinal disorders) | 41 | 13
Dyspepsia (Gastrointestinal disorders) | 99 | 11
Nausea (Gastrointestinal disorders) | 240 | 68
Stomatitis (Gastrointestinal disorders) | 81 | 11
Vomiting (Gastrointestinal disorders) | 189 | 39
Asthenia (General disorders) | 153 | 41
Fatigue (General disorders) | 202 | 69
Mucosal inflammation (General disorders) | 118 | 14
Oedema peripheral (General disorders) | 63 | 23
Pain (General disorders) | 49 | 24
Pyrexia (General disorders) | 57 | 12
Urinary tract infection (Infections and infestations) | 51 | 12
Aspartate aminotransferase increased (Investigations) | 29 | 6
Blood alkaline phosphatase increased (Investigations) | 37 | 17
Haemoglobin decreased (Investigations) | 36 | 6
Weight decreased (Investigations) | 115 | 25
Decreased appetite (Metabolism and nutrition disorders) | 237 | 52
Dehydration (Metabolism and nutrition disorders) | 32 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 35 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 56 | 26
Back pain (Musculoskeletal and connective tissue disorders) | 87 | 58
Bone pain (Musculoskeletal and connective tissue disorders) | 62 | 45
Muscle spasms (Musculoskeletal and connective tissue disorders) | 21 | 16
Muscular weakness (Musculoskeletal and connective tissue disorders) | 32 | 13
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 37 | 14
Pain in extremity (Musculoskeletal and connective tissue disorders) | 75 | 38
Dizziness (Nervous system disorders) | 49 | 16
Dysgeusia (Nervous system disorders) | 170 | 27
Headache (Nervous system disorders) | 50 | 17
Insomnia (Psychiatric disorders) | 40 | 19
Haematuria (Renal and urinary disorders) | 46 | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 46 | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 71 | 18
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 57 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 60 | 18
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 172 | 8
Petechiae (Skin and subcutaneous tissue disorders) | 41 | 4
Rash (Skin and subcutaneous tissue disorders) | 51 | 17
Skin discolouration (Skin and subcutaneous tissue disorders) | 33 | 4
Yellow skin (Skin and subcutaneous tissue disorders) | 78 | 6
Hypertension (Vascular disorders) | 150 | 17

LIMITATIONS AND CAVEATS:
A complete analysis was not performed due to the sponsors early termination of the clinical trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.